CLINICAL TRIAL: NCT00483808
Title: Renal Denervation in Patients With Refractory Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TP-015 & TP-038
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Denervation (Experimental): Renal denervation using the Symplicty Catheter
  Interventions: Device: Ardian Symplicity™ Catheter

INTERVENTIONS:
Device: Ardian Symplicity™ Catheter — Renal denervation using the Symplicity Catheter

SUMMARY:
To investigate the clinical utility of renal denervation in the treatment of refractory hypertension.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age.
* a systolic blood pressure of 160 mmHg or greater.
* receiving and adhering to full doses of an appropriate antihypertensive drug regimen for a minimum of two weeks prior to screening.
* agrees to have the study procedure(s) performed and additional procedures and evaluations, including repeat phlebotomy, imaging, urine analyses, and clinical examination.
* competent and willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria:

* renal arterial abnormalities
* end stage renal disease requiring dialysis or renal transplant
* serum Cr > 3, or calculated GFR < 45 ml/min
* has experienced MI, unstable angina pectoris, or CVA with 6 months
* others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To provide confirmation that renal denervation is safe and feasible. | 3 years

SECONDARY OUTCOMES:
Evidence of renal denervation; indication of physiologic response; assessment of device performance. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS,PhD, Principal Investigator — The Alfred Hospital and Monash University, Melbourne, VIC, Australia; Robert Whitbourn, MBBS, FRACP, Principal Investigator — St. Vincent's Hospital, Fitzroy, VIC, Australia
Locations (3):
- Australia (2):
  - St. Vincent's Hospital, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- John Paul II Hospital, Krakow, Poland

REFERENCES:
- [Derived] Eikelis N, Hering D, Marusic P, Duval J, Hammond LJ, Walton AS, Lambert EA, Esler MD, Lambert GW, Schlaich MP. The Effect of Renal Denervation on Plasma Adipokine Profile in Patients with Treatment Resistant Hypertension. Front Physiol. 2017 May 30;8:369. doi: 10.3389/fphys.2017.00369. eCollection 2017. PMID 28611687
- [Derived] Krum H, Schlaich MP, Sobotka PA, Bohm M, Mahfoud F, Rocha-Singh K, Katholi R, Esler MD. Percutaneous renal denervation in patients with treatment-resistant hypertension: final 3-year report of the Symplicity HTN-1 study. Lancet. 2014 Feb 15;383(9917):622-9. doi: 10.1016/S0140-6736(13)62192-3. Epub 2013 Nov 7. PMID 24210779
- [Derived] Schlaich MP, Hering D, Sobotka PA, Krum H, Esler MD. Renal denervation in human hypertension: mechanisms, current findings, and future prospects. Curr Hypertens Rep. 2012 Jun;14(3):247-53. doi: 10.1007/s11906-012-0264-9. PMID 22457244
- [Derived] Witkowski A, Prejbisz A, Florczak E, Kadziela J, Sliwinski P, Bielen P, Michalowska I, Kabat M, Warchol E, Januszewicz M, Narkiewicz K, Somers VK, Sobotka PA, Januszewicz A. Effects of renal sympathetic denervation on blood pressure, sleep apnea course, and glycemic control in patients with resistant hypertension and sleep apnea. Hypertension. 2011 Oct;58(4):559-65. doi: 10.1161/HYPERTENSIONAHA.111.173799. Epub 2011 Aug 15. PMID 21844482
- [Derived] Hering D, Esler MD, Krum H, Mahfoud F, Bohm M, Sobotka PA, Schlaich MP. Recent advances in the treatment of hypertension. Expert Rev Cardiovasc Ther. 2011 Jun;9(6):729-44. doi: 10.1586/erc.11.71. PMID 21714604
- [Derived] Schlaich MP, Sobotka PA, Krum H, Whitbourn R, Walton A, Esler MD. Renal denervation as a therapeutic approach for hypertension: novel implications for an old concept. Hypertension. 2009 Dec;54(6):1195-201. doi: 10.1161/HYPERTENSIONAHA.109.138610. Epub 2009 Oct 12. No abstract available. PMID 19822798
- [Derived] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353